CLINICAL TRIAL: NCT01083849
Title: Long-Term Therapy Outcomes When Treating CKD-patients With Paricalcitol in German Clinical Practice (TOP Study)
Brief Title: Long-Term Therapy Outcomes When Treating Chronic Kidney Disease (CKD) Patients With Paricalcitol in German and Austrian Clinical Practice
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-681
Record Dates: First submitted 2010-02-25; First posted 2010-03-10 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Insufficiency; Secondary Hyperparathyroidism
Keywords: Observational study; Paricalcitol; Treatment of Hyperparathyroidism; Chronic kidney disease stage 3, 4 and 5 (CKD stage 3, 4 and 5); Chronic Kidney Disease; Zemplar; sHPT; Secondary
MeSH Terms: conditions — Renal Insufficiency; Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paricalcitol: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, received paricalcitol injection or capsules, on an on-label basis in an everyday setting. Participants were observed for 12 months.

SUMMARY:
The purpose of this study is to obtain data on the safety and effectiveness of Zemplar® (paricalcitol) injection and paricalcitol capsules in real-life clinical practice. Participants, who have been treated with paricalcitol in-label in an everyday setting, have been included into this study. A period of 12 months has been chosen in order to also obtain experience on the maintenance dose and treatment optimization with paricalcitol injection and paricalcitol capsules in long-term use.

DETAILED DESCRIPTION:
According to protocol amendment of 16 October 2010 Austria is participating in this study.

Paricalcitol injection (intravenous (IV) therapy) was approved in Germany in December 2004 and in Austria in June 2003 for the prevention and treatment of secondary hyperparathyroidism in participants needing dialysis. In April 2008 in Germany and in January 2008 in Austria, paricalcitol capsules (for oral use (p.o.)) were launched for the prevention and treatment of secondary hyperparathyroidism in individuals with Chronic Kidney Disease stage 3 - 5 (i.e., predialysis and dialysis), thus enabling early treatment of participants with chronic kidney disease before they reach the stage of requiring dialysis.

Postmarketing observational studies with a well-planned study design, defined study protocol and biometrical estimates are necessary for a more profound understanding of the effectiveness and adverse drug reactions, especially those that are unknown or rare.

Accordingly, the purpose of this study is to obtain data on the safety and effectiveness of paricalcitol injection and capsules in real-life clinical practice. In this study, paricalcitol will be prescribed on an on-label basis in an everyday setting. A period of 12 months has been consciously chosen in order to also obtain experience on the maintenance dose and treatment optimization with paricalcitol injection and paricalcitol capsules in long-term use.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are based on the Summary of Product Characteristics for paricalcitol injection and capsules: Prevention and therapy of secondary hyperparathyroidism in the presence of chronic kidney disease
* Patients not treated with paricalcitol for at least 6 months prior to inclusion in this study

Exclusion Criteria:

* The contraindications listed in the Summary of Product Characteristics for paricalcitol injection and capsules apply
* An additional exclusion criterion is a parathyroid hormone- value of > 1000 pg/mL (which may be a sign of tertiary hyperparathyroidism) and existing treatment with paricalcitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating sites were facilities specialized in the treatment of chronic kidney disease and offices of community-based specialists/nephrologists in Germany and Austria.
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2008-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Decker-Burgard, MD, Study Director — AbbVie
Locations (87):
- Austria (11):
  - Site Reference ID/Investigator# 64522, Feldkirch
  - Site Reference ID/Investigator# 53506, Graz
  - Site Reference ID/Investigator# 53524, Graz
  - Site Reference ID/Investigator# 74733, Innsbruck
  - Site Reference ID/Investigator# 64523, Rottenmann
  - Site Reference ID/Investigator# 53525, Salzburg
  - Site Reference ID/Investigator# 53526, Sankt Pölten
  - Site Reference ID/Investigator# 69662, Steyr
  - Site Reference ID/Investigator# 53508, Vienna
  - Site Reference ID/Investigator# 53523, Vienna
  - Site Reference ID/Investigator# 53507, Vienna
- Germany (76):
  - Site Reference ID/Investigator# 28352, Aachen
  - Site Reference ID/Investigator# 28359, Alsfeld
  - Site Reference ID/Investigator# 28305, Arnstadt
  - Site Reference ID/Investigator# 28306, Aschersleben
  - Site Reference ID/Investigator# 28003, Augsburg
  - Site Reference ID/Investigator# 81613, Aurich
  - Site Reference ID/Investigator# 28017, Bad Bevensen
  - Site Reference ID/Investigator# 28301, Bad Nenndorf
  - Site Reference ID/Investigator# 28296, Balingen
  - Site Reference ID/Investigator# 28021, Berlin
  - Site Reference ID/Investigator# 28024, Berlin
  - Site Reference ID/Investigator# 28303, Berlin
  - Site Reference ID/Investigator# 54050, Berlin
  - Site Reference ID/Investigator# 28022, Bernburg
  - Site Reference ID/Investigator# 30862, Betzdorf
  - Site Reference ID/Investigator# 28007, Bielefeld
  - Site Reference ID/Investigator# 28304, Burg
  - Site Reference ID/Investigator# 28014, Coburg
  - Site Reference ID/Investigator# 28023, Cottbus
  - Site Reference ID/Investigator# 28134, Demmin
  - Site Reference ID/Investigator# 28037, Dresden
  - Site Reference ID/Investigator# 43903, Dresden
  - Site Reference ID/Investigator# 99777, Elmshorn
  - Site Reference ID/Investigator# 28284, Elsenfeld
  - Site Reference ID/Investigator# 124118, Emden
  - Site Reference ID/Investigator# 54054, Emsdetten
  - Site Reference ID/Investigator# 48864, Erfurt
  - Site Reference ID/Investigator# 72343, Erkelenz
  - Site Reference ID/Investigator# 28029, Eschweiler
  - Site Reference ID/Investigator# 28287, Friedrichroda
  - Site Reference ID/Investigator# 28276, Gera
  - Site Reference ID/Investigator# 28351, Halle
  - Site Reference ID/Investigator# 28280, Hamburg
  - Site Reference ID/Investigator# 48865, Hanover
  - Site Reference ID/Investigator# 28300, Heilbronn
  - Site Reference ID/Investigator# 28011, Herford
  - Site Reference ID/Investigator# 124119, Herne
  - Site Reference ID/Investigator# 28019, Herzberg
  - Site Reference ID/Investigator# 28135, Hildesheim
  - Site Reference ID/Investigator# 28286, Hoyerswerda
  - Site Reference ID/Investigator# 28353, Ilfeld
  - Site Reference ID/Investigator# 28044, Jena
  - Site Reference ID/Investigator# 48863, Kiel
  - Site Reference ID/Investigator# 28013, Lahr
  - Site Reference ID/Investigator# 28025, Loerrach
  - Site Reference ID/Investigator# 28290, Ludwigslust
  - Site Reference ID/Investigator# 10982, Magdeburg
  - Site Reference ID/Investigator# 28291, Malente
  - Site Reference ID/Investigator# 28036, Mannheim
  - Site Reference ID/Investigator# 28302, Marburg
  - Site Reference ID/Investigator# 54051, Minden
  - Site Reference ID/Investigator# 99778, Munich
  - Site Reference ID/Investigator# 28278, Müllheim
  - Site Reference ID/Investigator# 99776, Neumünster
  - Site Reference ID/Investigator# 124120, Nordhorn
  - Site Reference ID/Investigator# 28275, Nordhorn
  - Site Reference ID/Investigator# 43904, Oberstdorf
  - Site Reference ID/Investigator# 28277, Osnabrück
  - Site Reference ID/Investigator# 28297, Peine
  - Site Reference ID/Investigator# 28307, Pirmasens
  - Site Reference ID/Investigator# 28295, Potsdam
  - Site Reference ID/Investigator# 28294, Quedlinburg
  - Site Reference ID/Investigator# 48862, Rendsburg
  - Site Reference ID/Investigator# 28042, Ribnitz-Damgarten
  - Site Reference ID/Investigator# 28282, Rostock
  - Site Reference ID/Investigator# 28033, Saint Wendel
  - Site Reference ID/Investigator# 54052, Stuttgart
  - Site Reference ID/Investigator# 28005, Stuttgart
  - Site Reference ID/Investigator# 28020, Viersen
  - Site Reference ID/Investigator# 28293, Villingen-Schwenningen
  - Site Reference ID/Investigator# 28018, Völklingen
  - Site Reference ID/Investigator# 28298, Weißenfels
  - Site Reference ID/Investigator# 28292, Wetzlar
  - Site Reference ID/Investigator# 48882, Wiesbaden
  - Site Reference ID/Investigator# 28299, Wolfenbüttel
  - Site Reference ID/Investigator# 28279, Zwickau

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 761 participants were enrolled in the study, but two participants lacked information necessary for assignment to one of the analysis groups (pre-dialysis or dialysis). Hence, analysis was conducted with 759 participants.
Groups:
- Paricalcitol Pre-dialysis Group: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, and who were not yet on dialysis received paricalcitol injection or capsules, on an on-label basis in an everyday setting. Participants were observed for 12 months.
- Paricalcitol Dialysis Group: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, and on dialysis received paricalcitol injection or capsules, on an on-label basis in an everyday setting. Participants were observed for 12 months.
Period: Overall Study
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Started | 121 | 638
Completed | 61 | 527
Not Completed | 60 | 111

BASELINE CHARACTERISTICS:
Population: A total of 761 participants were enrolled in the study, however 2 participants lacked information necessary for assignment to one of the analysis groups. Hence, analysis was conducted with 759 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group | Total
Number analyzed (Participants) | 121 | 638 | 759
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (13.9) | 62.5 (14.9) | 62.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 291 | 338
  Male | 74 | 347 | 421
Duration of Chronic Kidney Disease [Mean (Standard Deviation); unit: months] — Duration of Chronic Kidney Disease until the start of the study
  months | 39.3 (36.0) | 71.2 (61.1) | 67.5 (59.6)
Duration of Secondary Hyperparathyroidism [Mean (Standard Deviation); unit: months] — Duration of Secondary Hyperparathyroidism until the start of the study
  months | 17.7 (20.6) | 43.9 (36.6) | 39.5 (35.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Intact Parathyroid Hormone (iPTH) Levels Within the Target Range After 12 Months
Description: Participants achieved Intact Parathyroid Hormone (iPTH) levels within the target range of Kidney Disease Quality Outcome Initiative (K/DOQI) treatment guidelines (Chronic Kidney Disease (CKD), stage 3: 35 to 70 pg/mL; CKD stage 4: 70 to 110 pg/mL; CKD stage 5: 150 to 300 pg/mL).
Time Frame: Up to 12 Months
Population: Participants with a determined chronic kidney disease (CKD) stage
Measure: Number; unit: percentage of participants
Groups:
- Paricalcitol: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, not treated with paricalcitol for at least 6 months prior inclusion in this study, received paricalcitol injection or capsules, on an on-label basis in an everyday setting. Participants were observed for 12 months.
Arm/Group | Paricalcitol
Number analyzed (Participants) | 718
percentage of participants
  Stage 3 [N=56] | 30.4
  Stage 4 [N=82] | 30.5
  Stage 5 [N=580] | 70.2

2. Secondary Outcome: Number of Participants With Hypercalcemia
Description: Hypercalcemia was defined as having a serum calcium level greater than 11.2 mg/dL (2.79 mmol/L), in one measurement. Serum calcium was measured at every study visit.
Time Frame: Months 0, 3, 6, 9, and 12
Population: The Pre-Dialysis and Dialysis groups were split into subgroups. Secondary endpoint investigations were done for the 733 participants in these Pre-Dialysis or Dialysis subgroups; 26 out of the 759 participants had a missing subgroup allocation.
Measure: Number; unit: participants
Groups:
- Paricalcitol Pre-dialysis Group: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, and who were not yet on dialysis received paricalcitol injection or capsules, prescribed on an on-label basis in an everyday setting. Participants were observed for 12 months.
- Paricalcitol Dialysis Group: Participants with chronic kidney disease and a diagnosis of secondary hyperparathyroidism, and on dialysis received paricalcitol injection or capsules, prescribed on an on-label basis in an everyday setting. Participants were observed for 12 months.
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
participants
  Month 0 | 1 | 2
  Month 3 | 2 | 6
  Month 6 | 1 | 4
  Month 9 | 1 | 4
  Month 12 | 1 | 5

3. Secondary Outcome: Number of Participants With Hyperphosphatemia
Description: Hyperphosphatemia was defined as having a serum phosphate level greater than 6.5 mg/dL (2.10 mmol/L), in one measurement. Serum phosphate was measured at every study visit.
Time Frame: Months 0, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
participants
  Month 0 | 5 | 192
  Month 3 | 8 | 153
  Month 6 | 8 | 151
  Month 9 | 9 | 133
  Month 12 | 8 | 128

4. Secondary Outcome: Number of Participants With Elevated Calcium-Phosphorus Product
Description: Elevated Calcium-Phosphorus Product was defined as having a calcium-phosphate product level greater than 65 mg^2/dL^2, in one measurement. Serum calcium-phosphorus product was measured at every study visit.
Time Frame: Months 0, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
participants
  Month 0 | 5 | 102
  Month 3 | 6 | 97
  Month 6 | 7 | 101
  Month 9 | 6 | 89
  Month 12 | 4 | 78

5. Secondary Outcome: Mean Duration of Hospitalization by Visit
Time Frame: Months 0, 3, 6, 9, and 11
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
days
  Month 0 | 1.3 (4.9) | 0.7 (4.0)
  Month 3 | 1.8 (4.4) | 0.8 (3.5)
  Month 6 | 2.9 (5.9) | 0.8 (4.3)
  Month 9 | 0.0 (0.0) | 0.8 (3.5)
  Month 11 | 0.9 (4.0) | 0.6 (3.9)

6. Secondary Outcome: Mean Duration of Disability by Visit
Time Frame: Months 0, 3, 6, 9, and 11
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
days
  Month 0 | 0.0 (0.0) | 0.3 (3.0)
  Month 3 | 4.7 (8.1) | 0.2 (2.0)
  Month 6 | 0.0 (0.0) | 0.4 (3.5)
  Month 9 | 0.0 (0.0) | 0.4 (3.1)
  Month 11 | 0.3 (1.0) | 0.4 (3.2)

7. Primary Outcome: Time to Achieve Target Range of Intact Parathyroid Hormone (iPTH) Levels Within the Target Range After 12 Months
Description: as for outcome 1
Time Frame: Up to 12 months
Population: Participants with a determined chronic kidney disease (CKD) stage
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Paricalcitol
Number analyzed (Participants) | 718
days
  Stage 3 [N=17] | 212.4 (203.93)
  Stage 4 [N=25] | 195.5 (118.3)
  Stage 5 [N=407] | 145.7 (107.1)

8. Secondary Outcome: Mean Intact Parathormone (iPTH) Levels by Visit
Time Frame: Months 0, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
pmol/L
  Month 0 | 29.65 (26.95) | 54.85 (29.51)
  Month 3 | 26.95 (36.94) | 37.20 (28.35)
  Month 6 | 23.01 (27.32) | 37.18 (30.08)
  Month 9 | 27.85 (33.95) | 36.54 (29.42)
  Month 12 | 29.57 (31.28) | 38.24 (33.76)

9. Secondary Outcome: Mean Calcium-Phosphate Product Levels by Visit
Time Frame: Months 0, 3, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol²/l²
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Number analyzed (Participants) | 96 | 637
mmol²/l²
  Month 0 | 3.32 (3.12) | 4.12 (1.29)
  Month 3 | 3.50 (1.46) | 4.30 (1.26)
  Month 6 | 3.62 (1.61) | 4.32 (1.22)
  Month 9 | 3.61 (1.37) | 4.25 (1.29)
  Month 12 | 3.48 (1.20) | 4.21 (1.31)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) occurring during the 12-month observation period from the date of initiation of paricalcitol treatment plus 30 days after the end of that period had to be recorded.
Description: Adverse Event investigations were done for the 733 participants which were in the predialysis (N=96) or dialysis subgroups (N=637).
Arm/Group | Paricalcitol Pre-dialysis Group | Paricalcitol Dialysis Group
Serious Adverse Events (participants affected / at risk) | 16/96 | 186/637
Other Adverse Events (participants affected / at risk) | 0/96 | 0/637
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol Pre-dialysis Group (N=96) | Paricalcitol Dialysis Group (N=637)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 3
Cardiac failure (Cardiac disorders) | 0 | 5
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 3
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 4
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticular hernia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 2
Death (General disorders) | 1 | 13
Device dislocation (General disorders) | 0 | 3
Device malfunction (General disorders) | 0 | 2
Device occlusion (General disorders) | 0 | 1
Fat necrosis (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Hernia obstructive (General disorders) | 0 | 1
Hyperplasia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 0 | 3
Sudden death (General disorders) | 0 | 1
Ulcer (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Device related sepsis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 2
Intervertebral discitis (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 4
Sepsis (Infections and infestations) | 0 | 8
Sinusitis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 3
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 2
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 12
Shunt stenosis (Injury, poisoning and procedural complications) | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 2
Angiogram (Investigations) | 0 | 1
Arteriogram coronary (Investigations) | 0 | 1
Blood parathyroid hormone increased (Investigations) | 0 | 1
Catheterisation cardiac (Investigations) | 0 | 2
Colonoscopy (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Endoscopy (Investigations) | 0 | 1
Endoscopy upper gastrointestinal tract (Investigations) | 0 | 2
Investigation (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
IIIrd nerve paresis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Abscess management (Surgical and medical procedures) | 0 | 1
Angioplasty (Surgical and medical procedures) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 8
Arteriovenous shunt operation (Surgical and medical procedures) | 1 | 3
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 1
Cataract operation (Surgical and medical procedures) | 0 | 1
Catheter placement (Surgical and medical procedures) | 1 | 1
Central venous catheterisation (Surgical and medical procedures) | 0 | 3
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Dialysis (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 7
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Leg amputation (Surgical and medical procedures) | 0 | 3
Mitral valve repair (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
Parathyroid gland operation (Surgical and medical procedures) | 0 | 1
Parathyroidectomy (Surgical and medical procedures) | 0 | 2
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1
Removal of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 | 1
Renal transplant (Surgical and medical procedures) | 0 | 3
Resection of rectum (Surgical and medical procedures) | 0 | 1
Stent placement (Surgical and medical procedures) | 0 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 3
Toe amputation (Surgical and medical procedures) | 0 | 2
Transplant (Surgical and medical procedures) | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 0 | 1
Urinary tract operation (Surgical and medical procedures) | 0 | 1
Venous operation (Surgical and medical procedures) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 2
Extremity necrosis (Vascular disorders) | 0 | 3
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 8
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 9
Poor peripheral circulation (Vascular disorders) | 0 | 1
Steal syndrome (Vascular disorders) | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.